CLINICAL TRIAL: NCT03822039
Title: Compliance Levels With WHO Checklist-based Infection Prevention Guidelines and Associated Surgical Site Infection Following Caesarean Delivery in Mulago Hospital
Brief Title: WHO Checklist- Based Infection Prevention Guidelines in Mulago Hospital
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Makerere University (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-085
Record Dates: First submitted 2018-09-11; First posted 2019-01-30 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2018-09

CONDITIONS: Surgical Site Infection
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This prospective cohort study will assess all mothers undergoing elective and emergency caesarean delivery in the labour ward theatre at Mulago National Referral Hospital based temporarily at Kawempe Hospital. Mothers will be recruited into the study systematically over a period of 3 months and follow-up daily until discharge or 30 days .

DETAILED DESCRIPTION:
To determine the level of compliance with WHO checklist-based infection prevention guidelines following caesarean delivery in Mulago National Referral Hospital, Kawempe.

To determine the association between compliance with WHO checklist-based infection prevention guidelines and surgical site infection following caesarean delivery in Mulago Hospital, Kawempe.

This prospective cohort study will assess all mothers undergoing elective and emergency caesarean delivery in the labour ward theatre at Mulago National Referral Hospital based temporarily at Kawempe Hospital. Mothers will be recruited into the study systematically over a period of 3 months and follow-up daily until discharge or 30 days of in-hospital stay for the purpose of documentation of surgical site infection. Data will be collected using the checklist expansion for antisepsis and infection control questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Mothers undergoing elective and emergency caesarean deliveries in Mulago National Referral Hospital, Kawempe in labour suite and gynaecology theatre.

Exclusion Criteria:

* Patient who is unconscious and unknown patient

Min Age: 15 Years | Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: Mothers undergoing Caesarean Deliveries in Mulago National Referral Hospital, Kawempe labour suite and gynaecology theatre.
Sampling Method: Probability Sample
Enrollment: 768 (Estimated)
Dates: Start 2018-07-16 (Actual); Primary Completion 2019-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Level of compliance with WHO checklist-based infection prevention guidelines following caesarean delivery among health care workers in Mulago Hospital, Kawempe | 24Hours
  Using a tool of 12 parameters from the WHO Surgical Safety Checklist-based infection prevention standards, each of the parameters will be given a score of 1 if it was obeyed by the respondent and a score of 0 if it was omitted. Compliance will be then expressed as a percentage completion of the items comprising the checklist.

SECONDARY OUTCOMES:
surgical site infection within 30 days of operation | 30 days
  Patients will be directly followed up during ward rounds until discharge and thereafter, telephone calls will be used every four days to enquire for development of surgical site infections such as fever, foul-smelling wound, redness around the incision, swelling/ induration at the wound site, burst wound.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Mbiya, Mbchb, Principal Investigator — Makerere University
Locations (1):
- Mulago hospital, Kampala, Mulago Hospital, Uganda

IPD SHARING:
Plan to Share IPD: No